CLINICAL TRIAL: NCT01661920
Title: Suitability of Antibiotic Treatment for Community-acquired Pneumonia
Brief Title: Suitability of Antibiotic Treatment for CAP
Acronym: CAPTIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, ALBERTO CAPELASTEGUI SAIZ, Head of Pneumology Service of Galdakao Hospital. PhD, MD., Hospital Galdakao-Usansolo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAPTIME; 2011-001067-51 (EudraCT Number)
Record Dates: First submitted 2012-07-26; First posted 2012-08-10 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Community Acquired Pneumonia
Keywords: Community Acquired Pneumonia.; Treatment duration
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- INTERVENTION GROUP (Experimental): Patients with diagnosis of CAP with shorten treatment, defined as 5 days antibiotic treatment.
  Interventions: Other: Intervention group
- CONTROL GROUP (Active Comparator): Patients with diagnosis of CAP which antibiotic treatment duration will be not modified by their doctors.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — Shorten the duration of antibiotic treatment from 7-10 days to 5 days.
  Arms: INTERVENTION GROUP
Other: Control group — Those antibiotic duration treatments which are not modified by their doctors.
  Arms: CONTROL GROUP

SUMMARY:
The duration of antibiotic treatment in community-acquired pneumonia (CAP) lasts about 9-10 days, and is determined empirically. The last North American guideline for CAP recommends using clinical stability criteria as a reference to establish the duration of antibiotic treatment, which would result in about 5 days of antibiotic use for the majority of pneumonia cases. In order to validate this proposal we propose to carry out a randomized multicenter double-blind (until the 5th day) clinical trial with adult CAP patients admitted to 4 hospitals in Euskadi. A control group (with routine treatment) will be compared with an intervention group (antibiotic treatment for at least 5 days, which will be interrupted if temperature is =< 37,8ºC for at least 48 hours and no more than one sign of clinical instability is assessed), with regards to: mortality at 15 days, clinical recovery by days 10 and 30, clinical improvement after days 5 and 10 as evaluated by PRO scales, duration of antibiotic treatment. A non-inferiority dichotomous sequential analysis will be performed (for mortality after 15 days, clinical recovery by day 10 and in follow-up at 30 days, clinical improvement after days 5 and 10, with PRO scales) as well as a superiority analysis for the duration of the antibiotic treatment. A total of 1100 patients will be recruited, following their signed consent, during the inclusion period (18 months). Stability criteria will be measured daily. The rest of the variables will be measured at admission and by telephone on days 10 and 30.

DETAILED DESCRIPTION:
Work hypothesis: We aim to carry out a comparative study between 2 groups of patients (control group, guideline group): in the control group the standard duration of antibiotic treatment will be applied; in the guideline group (intervention group) the duration of antibiotic treatment will be based upon the IDSA/ATS 2007 provisions (ref. 18), which are related to the time needed to reach clinical stability.

1. - Patients who follow the treatment protocol of the so-called control group, with routine treatment, in comparison to the clinical guideline group, will show similar results (sequential dichotomous non-inferiority analysis) in the following clinical parameters: A. Adverse results: 1st, mortality for any cause within the first 15 days after admission; 2nd, development of (major or minor) complications during the first 15 days after admission; B. Beneficial results: 1st, clinical recovery by the 10th day of treatment and in follow-up at 30 days; 2nd, clinical improvement on the 5th and 10th days of treatment, as evaluated by PRO scales.
2. - Patients who follow the treatment protocol of the so-called guideline group (intervention group), in comparison with the control group, with routine treatment, will show better results (superiority analysis) in the following parameters: c. Duration of antibiotic treatment as measured using 2 variables: 1.- the "duration of antibiotic treatment" after admission, expressed in days; 2.- "antibiotic-free days", defined as a period of at least 24 hours in which antibiotics are not given in the 30 day period after admission.

Goals: To validate the recommendations of the latest IDSA/ATS clinical guideline on duration of antibiotic treatment in pneumonia.

Main goals. To compare two treatment routines (control group with routine treatment vs clinical guideline group) based on results in the following clinical parameters:

A. Adverse results: 1st, mortality for any cause within the first 15 days after admission; 2nd, development of (major or minor) complications during the first 15 days after admission; B. Beneficial results: 1st, clinical recovery by the 10th day of treatment and in follow-up at 30 days; 2nd, clinical improvement on the 5th and 10th days of treatment, as evaluated by PRO scales.

2.- Patients who follow the treatment schema of the so-called guideline group (intervention group), in comparison with the control group, with routine treatment, will show better results (superiority analysis) in the following parameters: c. Duration of antibiotic treatment as measured using 2 variables: 1.- the "duration of antibiotic treatment" after admission, expressed in days; 2.- "antibiotic-free days", defined as a period of at least 24 hours in which antibiotics are not given in the 30 day period after admission.

Secondary goals: To compare a control group with routine treatment vs the clinical guideline group based on the following parameters:

1. In-hospital mortality for any cause. Mortality within 30 days after admission, whether related or unrelated to pneumonia.
2. Readmission within 30 days after admission for reasons related or unrelated to pneumonia.
3. Duration of hospital stay.
4. Days to return to normal activity.
5. Recurrence of initial infection or superinfection with need for additional or alternative antibiotics, within 30 days after admission.

Study design - Population under study. Inclusion/exclusion criteria - Main and secondary variables - Data analysis - Ethical and legal aspects (BCP compliance, insurance…) - Aspects related to the research medication (manufacturing, labeling, distribution…) - Funding sources of the medication Randomized multicenter double-blind (until the 5th day) clinical trial involving adult PAC patients (≥18 years of age) admitted to 4 teaching hospitals in Euskadi. All CAP patients hospitalized within a period of 18 months (October-April) will be evaluated for their eligibility. The study involves an intervention and will be undertaken in 2 parallel groups, where the duration of antibiotic treatment following routine clinical practice (control group) will be compared with its duration under the IDSA/ATS provisions for CAP (ref. 18) ("clinical guideline" group). Patients will be randomly assigned to the control group or the "clinical guideline" group on the third day of their hospital stay. Researchers will not be notified of the random assignment until day 5. In the control group patients will be treated according to routine practice for 9 days or longer. In this group there is no interference with the duration of antibiotic treatment. In the "clinical guideline" group patents will receive antibiotics for a minimum of 5 days, antibiotics will be discontinued if temperature is at ≤ 37,8ºC for 48 hours and no more than one sign of clinical instability (see section on definitions) is attested. Once this situation of stability is attained, at each of the participating hospitals a research team doctor will instruct the physician in charge of each patient to drop antibiotic treatment from that moment on.

In patients of the "clinical guideline" group the degree of compliance with the study algorythm will be noted and the reasons that justify skipping it if the case presents itself. The evolution of the clinical trial will be monitored by an independent monitoring team.

Research team members will not be involved in decisions related to discharge from the hospital. After hospital discharge all patient care will depend on the correspoding family physicians. A control visit will be scheduled for the 30th day after admission.

Study location. Multicenter study that will take place in 4 public network Bizkaian hospitals: Galdakao-Usansolo Hospital, Basurto Hospital, Txagorritxu Hospital and San Eloy Hospital.

Study subjects. For a period of 18 months all adult patients, 18 or older, admitted with CAP will be included sequentially. Pneumonia is defined as pulmonary infiltrate shown in a thoracic X-ray not known to be old, plus symptoms consistent with pneumonia, such as cough, dysnea, fever and/or pleuritic chest pain. The following patients will be excluded: patients with human immunodeficiency virus infection, immunosupressed patients (with a solid organ transplant, spelenectomy, treated with a prednisone dose of 10 mg/day or equivalent for longer than 30 days or with other immunodepressors, with neutropenia), those hospitalized in the 14 days prior and those living in assisted care facilities. Pneumonia cases caused by infrequent agents (i.e. P. aerouginosa, S. Aureus) will also be excluded, as well as infectious processes requiring an extended treatment with antibiotocs (i.e. bacterial endocarditis, abscesses), pneumonia cases with pleural effusion requiring a drainage tube, patients who were deceased or admitted to ICU before randomization and those not giving their informed consent.

A total of 1100 cases will be included during the period of study. Losses: those cases not registering the data corresponding to the main goals (loss estimate <5%). A comparative analysis between lost and non-lost patients. For that purpose socio-demographic and clinical variables will be included, as well as those related to severity at admission and the Charlson index (Charlson ME et al. J Chronic Dis 1987;40:373-83).

Ethical aspects. All patients will be informed about the study and they will be asked to give their informed consent (see annex 2). All data will be treated following the law for the protection of personal data (Organic Law 15/1999, 13-12). The study database will be protected with security access measures and the patients' identification data will stay separate from the rest of the information included in the database.

Sample size. We have chosen the equivalence hypothesis in mortality rates between the control group (with conventional guideline) and the intervention group ("clinical guideline group", with treatment template following clinical guideline recommendations). For a unilateral (non-inferiority) contrast (a=0.05, 1- b=0.80) 545 patients will be needed for each group, so as to be able to reject the null hypothesis of non-equivalence of the treatment following the new clinical guidelines as opposed to conventional guidelines. We have assumed an equivalence margin of 1% (http://people.ucalgary.ca/~patten/blackwelder.html). Sample size has been calculated assuming a 5% rate of losses during follow-up.

Independent variables. 1- severity at admission time. During the 24 hours following arrival at the hospital's Emergency Service the requisite variables will be gathered so as to calculate risk class as established by the Pneumonia Severity Index (PSI) (Fine MJ, et al. N Engl J Med 1997;36:243-50) and the CURB65 scale (Confusion, Urea nitrogen, Respiratory rate, Blood pressure, Age) (Lim WS, et al. Thorax 2003;58:377-82); 2- comorbidities; 3-Charlson index; 4- treatment given: antibiotic prior to admission; adherence of antibiotic treatment to SEPAR provisions; initiation of antibiotic treatment in the first 8 hours; transition from intravenous to oral medication; use of non-invasive mechanical ventilation; 5- bacteriological diagnosis. During the acute phase two hemocultures, a sputum culture and urinary antigen tests will be included, while blood tests for atypical bacteria will be performed during the acute and remission phases.

Dependent variables. 1- mortality for any cause in a 15 day period after admission. The in-hospital mortality and at 30 days will also be analyzed. 2- clinical recovery on the 10th (recovery test - see definitions section) and 30th days; 3- clinical evolution on the 5th and 10th treatment days, measured by PRO scales; a specific validated 18-item questionnaire will be used (Lamping DL, et al. Chest 2002;122:920-9); 4- duration of antibiotic treatment after the time of hospitalization (in days) and days without antibiotic (periods of 24 hours without antibiotic) until the 30th day. 5- hospital readmission within 30 days. 6- duration of hospital stay. 7- clinical recovery (number of days); 8- recurrence of the initial infection or superinfection with need for additional or alternative antibiotic treatment (within 30 days); 9- number of days off work due to disease (within 30 days); 10- number of days with adverse effects from the medication (within 30 days); 11- number of days with the usual (recreation or work) activity restricted by pneumonia (within 30 days); 12- in-hospital complications and at 30 days; 13- need for additional medication.

Information collection. Patients will be included in the study once they are admitted with PAC. A protocol for data collection in both study groups will be designed. Clinical stability criteria will be collected daily twice a day during the admission period. The other study variables will be collected during hospital stay and by means of a structured telephone interview on the 10th (unless the patient is still hospitalized) and 30th days. All the data will be collected by trained blinded staff.

Antibiotic treatment. All patients shall be treated according to SEPAR recommendations (Arch Bronconeumol 2010;46:543-58): group inpatients, not in ICU. Intravenous beta-lactam (amoxicillin/clavulanate or cefotaxime or ceftriasone) plus intravenous macrolide (azitromicyn or claritromicyn), or intravenous levofloxacine; group ICU-admitted patients. Intravenous beta-lactam (cefotaxime or ceftriasone) plus intravenous macrolide (azitromycin or claritromycin), or intravenous beta-lactam (cefotaxime or ceftriasone) plus intravenous levofloxacine. The Research Team will insist on starting antibiotic treatment as soon as possible and on patients being treated with fluoroquinolone or beta-lactam with macrolides. The ultimate decision corresponds to the physician in charge of the patient.

Definitions. Clinical instability: systolic arterial pressure <90 mmHg; breathing rate > 24 breath/min; heart rate >100 heartbeats/min; O2 saturation <90% or O2 arterial pressure <60mmHg. Patients receiving oxygen supplement will be considered stable with O2 ≥95% saturation. Clinical recovery (cure test): resolution or improvement of symptoms and clinical signs related to pneumonia without a need for additional or alternative antibiotic treatment. Clinical recovery on follow-up at 30 days: when there is a continuance of resolution or improvement of symptoms and clinical signs related to pneumonia without a need for additional or alternative antibiotic treatment. Recurrence: new (or worsening) symptoms and signs related to pneumonia and with a new infection of the respiratory tract in a patient considered cured on the 10th day visit.

Statistical analysis: For the descriptive analysis we will use averages, standard deviations, medians and ranks for the quantitave variables and percentages for the qualitative ones. The fundamental analyses will include: 1) first, and in order to make sure that randomization has been done correctly, the fundamental basal variables of the study will be compared between the intervention group and the control group to verify that there are no statistically significant differences between both groups in those variables. Intermediate analyses will be performed every three months of follow-up to see whether there are differences between both groups that may justify discontinuing the study. 2) To respond to the fundamental goals and hypotheses of the study univariate analyses will be performed comparing all the main and secondary dependent variables between the two groups of patients (main independent variable). A subanalysis with the most severe patients will also be conducted (PSI IV and V).

For the comparison of the quantitative variables between the control group and the intervention group Student's t test or Wilcoxon's non-parametric test will be used, depending on whether the studied variable follows a normal distribution or not. For the comparison of the qualitative variables a Chi-square test or Fisher's exact test will be used. In adition a comparative analysis of the basal characteristics of the lost and non-lost patients will be performed, using the same statistical tests previously mentioned.

Problems and Limitations of the Study: 1- As in every clinical trial, the main problem may be our patients' lack of interest to become a part of our study, although we will attempt to reduce the impact of this factor by explaining the study objectives, with its possible benefits and risks and its general interest, both for them and for the rest of pneumonia patients; 2- In the "clinical guideline" group the ultimate decision to discontinue antibiotic treatment after reaching clinical stability criteria will depend on the physician in charge of each patient. It is possible we may find occasional resistance to conform with the established protocol. In order to neutralize protocol transgressions as much as possible, the decision to discontinue antibiotic treatment will be analyzed previously at each hospital by a member of the research team, who will relay it to the physician in charge. This way we will on the one hand ensure the compliance of each case to what is established in the clinical trial, and on the other, encourage the individual physician's cooperation. At any rate, if the protocol is skipped, the reasons surrounding the case will be recorded. 3- Multicenter studies are complicated from an operational point of view. There is the possibility that the ratio between eligible and included patients might differ from one location to the other(s), or that the number of cases included bears no relationship with the size of the service population. In order to neutralize this effect we will introduce the hospital factor in our statistical analyses, besides studying each hospital's caseload separately and comparing them all.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older,
* admitted with CAP will be included sequentially. Pneumonia is defined as pulmonary infiltrate shown in a thoracic X-ray not known to be old,

Exclusion Criteria:

* patients with human immunodeficiency virus infection,
* immunosupressed patients (with a solid organ transplant, spelenectomy, treated with a prednisone dose of 10 mg/day or equivalent for longer than 30 days or with other immunodepressors, with neutropenia),
* those hospitalized in the 14 days prior and those living in assisted care facilities.
* pneumonia cases caused by infrequent agents (i.e. P. aerouginosa, S. Aureus) will also be excluded, as well as infectious processes requiring an extended treatment with antibiotocs (i.e. bacterial endocarditis, abscesses),
* pneumonia cases with pleural effusion requiring a drainage tube,
* patients who were deceased or admitted to ICU before randomization and those not giving their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
duration of the antibiotic treatment | 30 days
  days taht the patient takes an antibiotic treatment, adding intravenous and oral
mortality | 15 days
  the mortality in fifteen days
clinical cure | 10 days
  resolution or improvement of symptoms and clinical signs related to pneumonia without a need for additional or alternative antibiotic treatment.
clinical cure | 30 days
  resolution or improvement of symptoms and clinical signs related to pneumonia without a need for additional or alternative antibiotic treatment.

SECONDARY OUTCOMES:
1- In-hospital mortality for any cause | 30 days
  Mortality within 30 days after admission, whether related or unrelated to pneumonia.
Readmission | 30 days
  Readmission within 30 days after admission for reasons related or unrelated to pneumonia.
Days needed to reach clinical stability | 30 days
  Days off work due to disease. Days with restricted regular activity (work or recreation) due to pneumonia. Days with adverse effects due to medication.
Recurrence | 30 days
  new (or worsening) symptoms and signs related to pneumonia and with a new infection of the respiratory tract in a patient considered cured on the 10th day visit.
Duration of hospital stay | 30 days
  days the patient needs to be hospitalized for pneumonia
days to return to normal activity | 30 days
  days the patient needs to carry out their daily lives

CONTACTS AND LOCATIONS:
Overall Officials: ALBERTO CAPELASTEGUI, PhD, MD, Principal Investigator — Osakidetza
Locations (4):
- Spain (4):
  - Hospital Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital San Eloy, Barakaldo, Bizkaia
  - Hospital Basurto, Bilbao, Bizkaia
  - Hospital Galdakao, Galdakao, Bizkaia

REFERENCES:
- [Result] File TM Jr. Clinical efficacy of newer agents in short-duration therapy for community-acquired pneumonia. Clin Infect Dis. 2004 Sep 1;39 Suppl 3:S159-64. doi: 10.1086/421354. PMID 15546111
- [Result] File TM Jr, Niederman MS. Antimicrobial therapy of community-acquired pneumonia. Infect Dis Clin North Am. 2004 Dec;18(4):993-1016, xi. doi: 10.1016/j.idc.2004.07.011. PMID 15555836
- [Result] Nicolau DP. Predicting antibacterial response from pharmacodynamic and pharmacokinetic profiles. Infection. 2001 Dec;29 Suppl 2:11-5. PMID 11785851
- [Result] Mandell LA, File TM Jr. Short-course treatment of community-acquired pneumonia. Clin Infect Dis. 2003 Sep 15;37(6):761-3. doi: 10.1086/377567. Epub 2003 Aug 28. No abstract available. PMID 12955635
- [Result] Durrington HJ, Summers C. Recent changes in the management of community acquired pneumonia in adults. BMJ. 2008 Jun 21;336(7658):1429-33. doi: 10.1136/bmj.a285. No abstract available. PMID 18566081
- [Result] Nobre V, Harbarth S, Graf JD, Rohner P, Pugin J. Use of procalcitonin to shorten antibiotic treatment duration in septic patients: a randomized trial. Am J Respir Crit Care Med. 2008 Mar 1;177(5):498-505. doi: 10.1164/rccm.200708-1238OC. Epub 2007 Dec 20. PMID 18096708
- [Result] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417
- [Result] Chastre J, Wolff M, Fagon JY, Chevret S, Thomas F, Wermert D, Clementi E, Gonzalez J, Jusserand D, Asfar P, Perrin D, Fieux F, Aubas S; PneumA Trial Group. Comparison of 8 vs 15 days of antibiotic therapy for ventilator-associated pneumonia in adults: a randomized trial. JAMA. 2003 Nov 19;290(19):2588-98. doi: 10.1001/jama.290.19.2588. PMID 14625336
- [Result] Montravers P, Fagon JY, Chastre J, Lecso M, Dombret MC, Trouillet JL, Gibert C. Follow-up protected specimen brushes to assess treatment in nosocomial pneumonia. Am Rev Respir Dis. 1993 Jan;147(1):38-44. doi: 10.1164/ajrccm/147.1.38. PMID 8420428
- [Result] Li JZ, Winston LG, Moore DH, Bent S. Efficacy of short-course antibiotic regimens for community-acquired pneumonia: a meta-analysis. Am J Med. 2007 Sep;120(9):783-90. doi: 10.1016/j.amjmed.2007.04.023. PMID 17765048
- [Result] el Moussaoui R, de Borgie CA, van den Broek P, Hustinx WN, Bresser P, van den Berk GE, Poley JW, van den Berg B, Krouwels FH, Bonten MJ, Weenink C, Bossuyt PM, Speelman P, Opmeer BC, Prins JM. Effectiveness of discontinuing antibiotic treatment after three days versus eight days in mild to moderate-severe community acquired pneumonia: randomised, double blind study. BMJ. 2006 Jun 10;332(7554):1355. doi: 10.1136/bmj.332.7554.1355. PMID 16763247
- [Result] Dunbar LM, Wunderink RG, Habib MP, Smith LG, Tennenberg AM, Khashab MM, Wiesinger BA, Xiang JX, Zadeikis N, Kahn JB. High-dose, short-course levofloxacin for community-acquired pneumonia: a new treatment paradigm. Clin Infect Dis. 2003 Sep 15;37(6):752-60. doi: 10.1086/377539. Epub 2003 Aug 28. PMID 12955634
- [Result] Slama TG, Amin A, Brunton SA, File TM Jr, Milkovich G, Rodvold KA, Sahm DF, Varon J, Weiland D Jr; Council for Appropriate and Rational Antibiotic Therapy (CARAT). A clinician's guide to the appropriate and accurate use of antibiotics: the Council for Appropriate and Rational Antibiotic Therapy (CARAT) criteria. Am J Med. 2005 Jul;118 Suppl 7A:1S-6S. doi: 10.1016/j.amjmed.2005.05.007. PMID 15993671
- [Result] Schrag SJ, Pena C, Fernandez J, Sanchez J, Gomez V, Perez E, Feris JM, Besser RE. Effect of short-course, high-dose amoxicillin therapy on resistant pneumococcal carriage: a randomized trial. JAMA. 2001 Jul 4;286(1):49-56. doi: 10.1001/jama.286.1.49. PMID 11434826
- [Result] Guillemot D, Carbon C, Balkau B, Geslin P, Lecoeur H, Vauzelle-Kervroedan F, Bouvenot G, Eschwege E. Low dosage and long treatment duration of beta-lactam: risk factors for carriage of penicillin-resistant Streptococcus pneumoniae. JAMA. 1998 Feb 4;279(5):365-70. doi: 10.1001/jama.279.5.365. PMID 9459469
- [Result] Kardas P. Patient compliance with antibiotic treatment for respiratory tract infections. J Antimicrob Chemother. 2002 Jun;49(6):897-903. doi: 10.1093/jac/dkf046. PMID 12039881
- [Result] Lim WS, Baudouin SV, George RC, Hill AT, Jamieson C, Le Jeune I, Macfarlane JT, Read RC, Roberts HJ, Levy ML, Wani M, Woodhead MA; Pneumonia Guidelines Committee of the BTS Standards of Care Committee. BTS guidelines for the management of community acquired pneumonia in adults: update 2009. Thorax. 2009 Oct;64 Suppl 3:iii1-55. doi: 10.1136/thx.2009.121434. No abstract available. PMID 19783532
- [Result] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Result] Halm EA, Fine MJ, Marrie TJ, Coley CM, Kapoor WN, Obrosky DS, Singer DE. Time to clinical stability in patients hospitalized with community-acquired pneumonia: implications for practice guidelines. JAMA. 1998 May 13;279(18):1452-7. doi: 10.1001/jama.279.18.1452. PMID 9600479
- [Result] Halm EA, Fine MJ, Kapoor WN, Singer DE, Marrie TJ, Siu AL. Instability on hospital discharge and the risk of adverse outcomes in patients with pneumonia. Arch Intern Med. 2002 Jun 10;162(11):1278-84. doi: 10.1001/archinte.162.11.1278. PMID 12038946
- [Result] Capelastegui A, Espana PP, Bilbao A, Martinez-Vazquez M, Gorordo I, Oribe M, Urrutia I, Quintana JM. Pneumonia: criteria for patient instability on hospital discharge. Chest. 2008 Sep;134(3):595-600. doi: 10.1378/chest.07-3039. Epub 2008 May 19. PMID 18490403
- [Result] Christ-Crain M, Muller B. Biomarkers in respiratory tract infections: diagnostic guides to antibiotic prescription, prognostic markers and mediators. Eur Respir J. 2007 Sep;30(3):556-73. doi: 10.1183/09031936.00166106. PMID 17766633
- [Result] Chalmers JD, Singanayagam A, Hill AT. C-reactive protein is an independent predictor of severity in community-acquired pneumonia. Am J Med. 2008 Mar;121(3):219-25. doi: 10.1016/j.amjmed.2007.10.033. PMID 18328306
- [Result] Menendez R, Cavalcanti M, Reyes S, Mensa J, Martinez R, Marcos MA, Filella X, Niederman M, Torres A. Markers of treatment failure in hospitalised community acquired pneumonia. Thorax. 2008 May;63(5):447-52. doi: 10.1136/thx.2007.086785. Epub 2008 Feb 1. PMID 18245147
- [Result] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- [Result] Schuetz P, Christ-Crain M, Thomann R, Falconnier C, Wolbers M, Widmer I, Neidert S, Fricker T, Blum C, Schild U, Regez K, Schoenenberger R, Henzen C, Bregenzer T, Hoess C, Krause M, Bucher HC, Zimmerli W, Mueller B; ProHOSP Study Group. Effect of procalcitonin-based guidelines vs standard guidelines on antibiotic use in lower respiratory tract infections: the ProHOSP randomized controlled trial. JAMA. 2009 Sep 9;302(10):1059-66. doi: 10.1001/jama.2009.1297. PMID 19738090